CLINICAL TRIAL: NCT04943718
Title: Personalized Vaccine for Patients With Recurrent Malignant Glioma: a Single-arm, Single-center, Open-labeled Study
Brief Title: Personalized Vaccine for Patients With Recurrent Malignant Glioma
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xuanwu Hospital, Beijing (Other)
Collaborators: Beijing Neoantigen Biotechnology Company (Unknown)
Responsible Party: Principal Investigator, Qingtang Lin, Director, glioma immunotherapy program, Xuanwu Hospital, Beijing
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2019-127
Record Dates: First submitted 2021-06-13; First posted 2021-06-29 (Actual); Last update posted 2021-06-29 (Actual); Status verified 2021-06

CONDITIONS: Malignant Glioma; Recurrent Glioma
MeSH Terms: conditions — Glioma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- personalized vaccine (Experimental): patients with recurrent malignant gliomas enrolled into this arm will receive the personalized vaccine through sub-cutaneous.
  Interventions: Biological: personalized vaccine

INTERVENTIONS:
Biological: personalized vaccine — Based on genetic and transcriptional sequencing information, personalized peptide vaccines would be designed and produced; patients would be vaccinated on day 1, 4, 8 ,15, 22 and then on week 12, 20.

SUMMARY:
A single-arm, single-center, open-labeled study will be conducted with an aim to investigate the feasibility, safety, and efficacy of the personalized vaccine for patients with recurrent malignant glioma.

ELIGIBILITY:
Inclusion Criteria:

* age 18-70;
* signed inform consent;
* patients with recurrent malignant glioma; have received surgery, radiotherapy, chemotherapy;
* patients' tumor tissue should have a high mutation load(>10 TMB); be genetically unstable; at least have 10 neoantigens;
* should be able to provide tumor tissue and peripheral blood for sequencing and flow cytometry analysis;
* at least three months post last operation; one month after the completion of the last anti-drug therapy or radiotherapy;
* have not received any immune therapy;
* at least have one measurable lesion;
* KPS >60;
* estimated survival > 3 months
* patients should have adequate organ and bone marrow function;

Exclusion Criteria:

* female patient is breastfeeding or pregnant;
* known history of allergy to peptides or other stimulating factors (i.e. GM-CSF);
* known history of Graft-Versus-Host Disease (GVHD);
* participation in gene therapy;
* other malignancy;
* systemic disease: i.e., severe infection; HIV;
* other conditions upon investigator's judgement;

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2021-07-15 (Estimated); Primary Completion 2023-06-13 (Estimated); Study Completion 2024-06-13 (Estimated)

PRIMARY OUTCOMES:
incidences of advent events and severe advent events | from initiation of study treatment to 28 weeks post-vaccination
  would be monitored and measured according to the National Cancer Institute Common Terminology Criteria for Adverse Events (version 4.X.)

SECONDARY OUTCOMES:
object response rate (ORR) according to iRANO criteria | from initiation of study treatment to 24 weeks post-vaccination (last shot)
  ORR including complete response (CR) and partial response (PR) would be assessed and measured based on the conditions proposed by iRANO criteria
progression free survival (PFS) | up to 48 weeks post-vaccination(last shot)
  time interval (measured in weeks) between initiation of study treatment to progression of disease
overall survival (OS) | up to 48 weeks post-vaccination(last shot)
  time interval (measured in weeks) from initiation of study treatment to the death of patients
immune response based on the criteria encoded by GRT-C903 and GRT-R904 | Baseline to end of treatment (up to approximately 12 months)
  humoral and cellular immune responses including generation of specific antibodies, inflammatory factors, immune cells, will be measured as proposed by GRT-C903 and GRT-R904

CONTACTS AND LOCATIONS:
Locations (1):
- Xuanwu Hospital, Capital Medical University, Beijing, Beijing Municipality, China